CLINICAL TRIAL: NCT01504061
Title: The Comparison of Mederma® N&I to Mederma® Ultra Gel to Reduce the Appearance of Post Surgical Scars
Brief Title: Mederma to Reduce Appearance of Post Surgical Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: MUS90025-4007-0
Record Dates: First submitted 2011-12-06; First posted 2012-01-05 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Scars
Keywords: surgical; scars; Mederma
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mederma Ultra Gel (Experimental)
  Interventions: Other: Mederma Ultra Gel
- Mederma N&I (Active Comparator)
  Interventions: Other: Mederma N&I

INTERVENTIONS:
Other: Mederma N&I — Topical gel applied three times a day for eight weeks.
  Arms: Mederma N&I
Other: Mederma Ultra Gel — Topical gel applied once daily for eight weeks.
  Arms: Mederma Ultra Gel

SUMMARY:
This is a single-center, 20-subject, investigator-blinded study to evaluate the effect of Mederma N&I to Mederma Ultra Gel on the appearance of post-surgical scars.

DETAILED DESCRIPTION:
This is a 10-week research study designed to compare the effect of two gels on the appearance of post surgical scarring of the chest and/or back. The subject will be asked to identify two symmetrical skin growths that they would like to have removed: one on the left chest and/or back and one on the right chest and/or back. Additionally, the subject will identify a third skin growth that they would like removed which is a reasonable distance from the two symmetrical skin growths and will be located either on the back or the chest.

Inclusion Criteria:

* Healthy male and non pregnant female subjects ≥18 years of age
* have seborrheic keratoses on the right and left chest and/or back

Exclusion Criteria:

-Subjects with known allergies or sensitivities to ingredients contained in the test product including onion extract and Lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18-70 years of age, of any race or sex.
* Subjects must be Fitzpatrick skin type I-VI.
* Subjects must have two symmetrical upper chest and/or back seborrheic keratoses and in the opinion of the investigator are good candidates for the study.

Exclusion Criteria:

* Subjects with known allergies or sensitivities to ingredients contained in the test product including onion extract and Lidocaine.
* Subjects with known history of keloids or hypertrophic scars.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Investigator assessment of post-surgical scar appearance (indices are erythema, softness, texture, and overall appearance). This assessment is accompanied by photography and dermaspectrophotometry. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Girish Munavalli, MD, MHS, Principal Investigator — Dermatology, Laser, and Vein Specialists of Carolinas, PLLC
Locations (1):
- Dermatology, Laser, and Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina, United States